CLINICAL TRIAL: NCT06760806
Title: Evaluation of Toxicities in Patients Treated With Palliative Radiotherapy at Policlinico Sant Orsola of Bologna - patieNts treAted wIth palliatiVe radiothErapy - NAIVE
Brief Title: Evaluation of Toxicities in Patients Treated With Palliative Radiotherapy at Policlinico Sant Orsola of Bologna.
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: NAIVE
Record Dates: First submitted 2024-12-01; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-09

CONDITIONS: Palliative Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to assess the outcome in palliative patients, particularly in terms of symptom resolution or alleviation, after radiation treatment of the various tumours analysed, in relation to the treatment setting, dosages and techniques used both for newly diagnosed tumours and for cases already diagnosed and treated at the Radiotherapy Unit of the Sant Orsola Hospital.

DETAILED DESCRIPTION:
Malignant neoplasms are frequent in the general population, particularly in countries with a high development index. In Europe, the incidence of malignant tumours in 2018 was almost 570 cases/100,000 inhabitants, while mortality in the same year was over 260 cases/100,000 inhabitants. In Italy, more than 175,000 new cancers were diagnosed in 2018, while the prevalence of malignant neoplasms in our country is 1990 cases/100,000 inhabitants. The therapy of neoplastic pathology is in most cases multimodal, and the various treatments can be adjuvant or neoadjuvant depending on the neoplasm treated and the strategy adopted from time to time. In addition, radiotherapy can play a key role in advanced disease, either with curative intent or with palliative intent on symptoms. Radiotherapy is one of the most effective means of providing palliation of cancer symptoms. The location of the symptom is essential to define a correct treatment plan, as the therapeutic approach will be different if the symptom is caused by the locally advanced primary tumour or by metastases. The symptoms most commonly relieved with palliative radiotherapy are pain, bleeding and obstruction.

Bone metastases are the most frequent cause of cancer-related pain and over 70% of patients with bone metastases are symptomatic. One of the most important goals in the treatment of bone metastases is to alleviate suffering and maintain an ability to manage daily activities. Radiotherapy plays a key role in improving the quality of life of these patients. Dosages, fractionations and techniques vary depending on the type of neoplasm treated, fractionations and techniques vary depending on the type of neoplasm treated, its location and the type of symptom to be palliated, as do the possible acute and late toxicities in relation to the characteristics of the treatment and, of course, the anatomical region irradiated. Systematic collection of data on palliative radiation treatment in different malignancies may make it possible to assess outcomes in relation to dosages, fractionation and techniques adopted in combination with other therapies, with the characteristics of the disease (bioprofile, histotype, stage, etc.) and of the patient (age, gender, comorbidities, etc...) The aim of the study is to evaluate the outcome in palliative patients, particularly in terms of symptom resolution or alleviation, after radiation treatment of the different tumours analysed, in relation to treatment setting, dosages and techniques used both for new neoplasm diagnoses and for cases already diagnosed and treated at the Radiatherapy Department of Sant Orsola Hospital.

The study is observational, retrospective and prospective, single-centre, spontaneous.

The structured collection of data necessary for the evaluation of the objectives will cover the period of observation period from 01/01/2000 to 31/12/2027.

ELIGIBILITY:
Inclusion Criteria:

* adult patients of either sex with a new or previous diagnosis of malignant neoplasm since 1st January 2000
* patients treated with paliative radiotherapy
* obtaining of informed consent

Exclusion Criteria:

* adult patients of either sex with a new or previous diagnosis of malignant neoplasm who choose not to undergo radiotherapy treatment
* patients enrolled in other studies
* pregnant or breastfeeding women

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Every patient with a neoplastic disease admitted to the radiotherapy department for palliative or follow-up radiation treatment.
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2021-01-21 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Symptom resolution or attenuation | From the start of therapy to the last follow-up at 12 months
  Evaluate the outcome in palliative patients, particularly in terms of symptom resolution or alleviation, after radiation treatment of the different tumours analysed, in relation to the treatment setting, dosages and techniques used

SECONDARY OUTCOMES:
Acute toxicity in relation to different radiotherapy disages and techniques and patient characteristics | immediate to 6 months after radiotherapy
  acute toxicity after radiotherapy, evaluated according to CTCAE v.5
Late toxicity in relation to different radiotherapy disages and techniques and patient characteristics | from 6 months after radiotherapy, through study completion, an average of 1 year
  late toxicity after completion of treatments, evaluated according to CTCAE v.5
Incidence of reprocessing and its characteristics | During follow ups through study completion, an average of 1 year
Symptom-free survival | During the follow-ups, up to the last one at 12 months
  Disease-free survival assessed based on the presence or absence of local, nodal, or metastatic recurrences
Overall survival | From enrollment to the last follow-up at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alessio Giuseppe Morganti, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero - Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No